CLINICAL TRIAL: NCT06921382
Title: Breastfeeding Intervention to Prevent Obesity Among Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Greensboro (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-FY24-392; R01DK140892 (NIH)
Record Dates: First submitted 2025-02-26; First posted 2025-04-10 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Breastfeeding Self-Efficacy; Breastfeeding Continuation; Breastfeeding Duration; Breastfeeding Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (peer counseling and funds) (Experimental): Participants in the intervention condition will be matched with Spanish-speaking peer counselors who will visit mothers at home regularly (weekly at the beginning of the study, monthly at the end of the study). In Month 1, mothers can choose to receive a $150 gift card or an electric breast pump. In Months 2-5, if infants are signed up for the WIC exclusive breastfeeding package, infants will receive $100 and mothers will receive $50. If infants are signed up for the WIC partial breastfeeding package, infants will receive $50 and mothers will receive $30.
  Interventions: Behavioral: Peer counseling; Behavioral: Additional funds
- Control group (No Intervention): Participants in the control condition will receive care-as-usual. For example, they will have access to WIC services, which can include peer counseling.

INTERVENTIONS:
Behavioral: Peer counseling — Participants in the intervention condition will be matched with Spanish-speaking peer counselors who will visit mothers at home regularly (weekly at the beginning of the study, monthly at the end of the study).
  Arms: Intervention group (peer counseling and funds)
Behavioral: Additional funds — In Month 1, mothers can choose to receive a $150 gift card or an electric breast pump. In Months 2-5, if infants are signed up for the WIC exclusive breastfeeding package, infants will receive $100 and mothers will receive $50. If infants are signed up for the WIC partial breastfeeding package, infants will receive $50 and mothers will receive $30.
  Arms: Intervention group (peer counseling and funds)

SUMMARY:
The goal of this clinical trial is to learn how to improve exclusive breastfeeding rates. The main questions it aims to answer are:

Do Hispanic mothers benefit from peer counseling support from peer counselors who can speak Spanish? Are mothers more likely to continue exclusive breastfeeding if additional funds are given so that the WIC exclusive breastfeeding package has the same cash value as the WIC formula feeding package?

Researchers will compare participants in the intervention group (who receive peer counseling and additional funds) to a control group (who do not receive peer counseling or additional funds) to see if the intervention package improves breastfeeding rates.

All participants (intervention and control) will complete weekly surveys about their feeding experiences ($8 per week). Members of the research team will also take infant weight/length measurements at home (twice during the first month and then at 2, 4, and 6 months). Participants will be recruited during pregnancy and the study will last for the first 6 months after their babies are born. Mothers and their infants are both participants in the study.

Participants in the intervention condition will also be matched with Spanish-speaking peer counselors who will visit mothers at home regularly (weekly at the beginning of the study, monthly at the end of the study). In Month 1, mothers can choose to receive a $150 gift card or an electric breast pump. In Months 2-5, if infants are signed up for the WIC exclusive breastfeeding package, infants will receive $100 and mothers will receive $50. If infants are signed up for the WIC partial breastfeeding package, infants will receive $50 and mothers will receive $30.

ELIGIBILITY:
Mothers and infants are both participants in the study. By the time study activities start, infants will be around 5 days old.

Inclusion Criteria Set 1 (determined at prenatal recruitment):

1. Confirmation of Hispanic origin
2. Receives or eligible for WIC
3. Mother is 18 years or older
4. Singleton pregnancy
5. Mother intends to breastfeed.

Inclusion Criteria Set 2 (determined after infants are born):

1. Infant gestational age 37 weeks or more
2. Normal infant birth weight (i.e., > 5 lbs 8 oz.)
3. Breastfeeding has been initiated
4. No congenital or other health issues (such as cleft palate) identified that require specific accommodations for feeding.

Exclusion Criteria:

1. Mothers below 18 years of age.
2. Mothers do not plan to breastfeed.
3. Mothers not eligible to participate in the WIC program due to high household income
4. Non-singleton pregnancy.

Min Age: 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Exclusive breastfeeding | From enrollment to the end of the study at 6 months
  Weeks of exclusive breastfeeding. Mothers will complete weekly surveys about their feeding experience.
Infant measurements | From enrollment to the end of the study at 6 months
  A member of the research team will take infant weight and length measurements at participants' homes. Measurements will be taken twice during the first month and then at the end of months 2, 4, and 6. Measurements will be converted into weight-for-age z-scores according to the World Health Organization Child Growth Standards (birth to 24 months). Scores typically range from about -6 to +6, with higher scores indicating greater length relative to age. A score of 0 represents the median for the reference population.

CONTACTS AND LOCATIONS:
Overall Officials: Jasmine M DeJesus, PhD, Principal Investigator — UNC Greensboro; Jigna M Dharod, PhD, Principal Investigator — UNC Greensboro; Aunchalee E. L. Palmquist, PhD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - WIC Guilford County, Greensboro, North Carolina
  - Cone Health, Greensboro, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided
It is critical to reassure participants that the investigators will not share their personal information, so it might not be possible to share individual participant data, even if it is de-identified.

REFERENCES:
- See also: Description on NIH reporter — https://reporter.nih.gov/search/ryyk6IFhmk6mc8_J90h2NQ/project-details/10944397